CLINICAL TRIAL: NCT00001298
Title: A Trial of Carboxypeptidase-G2 (CPDG2) and Thymidine for the Management of Patients With Methotrexate Toxicity and Renal Dysfunction
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 920134; 92-C-0134
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2000-02

CONDITIONS: Kidney Diseases
Keywords: Antibody; DAMPA; Enzyme; Kidney; Pharmacokinetics; Thymidine; Toxicity
MeSH Terms: conditions — Kidney Diseases | interventions — gamma-Glutamyl Hydrolase

INTERVENTIONS:
Drug: carboxypeptidase-G2

SUMMARY:
High dose methotrexate with leucovorin rescue has demonstrated activity in numerous malignancies. Although high dose methotrexate is generally well tolerated, unpredictable life-threatening toxicity can occur. For patients who have markedly delayed clearance of methotrexate secondary to renal dysfunction, therapeutic options are few and are of limited efficacy. Carboxypeptidase-G2 inactivates methotrexate by hydrolyzing its C-terminal glutamate residue. Carboxypeptidase-G2 could be used to rescue patients with renal dysfunction and delayed methotrexate excretion, as it provides an alternative to renal clearance as a route of elimination.

DETAILED DESCRIPTION:
High dose methotrexate with leucovorin rescue has demonstrated activity in numerous malignancies. Although high dose methotrexate is generally well tolerated, unpredictable life-threatening toxicity can occur. For patients who have markedly delayed clearance of methotrexate secondary to renal dysfunction, therapeutic options are few and are of limited efficacy. Carboxypeptidase-G2 inactivates methotrexate by hydrolyzing its C-terminal glutamate residue. Carboxypeptidase-G2 could be used to rescue patients with renal dysfunction and delayed methotrexate excretion, as it provides an alternative to renal clearance as a route of elimination.

ELIGIBILITY:
Patients of any age at risk for life-threatening toxicity following MTX administration secondary to delayed drug excretion as defined by:

Plasma MTX concentration at least 10 micromoles/liter more than 42 hours after the start of the MTX infusion; OR

Creatinine at least 1.5 times the upper limit of normal or creatinine clearance less than 60 ml/sqm/min and delayed MTX excretion documented by plasma MTX concentration measurements (at least 2 standard deviations above the mean) at least 12 hours following MTX administration.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10
Dates: Start 1992-03; Study Completion 2001-01

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Adamson PC, Balis FM, McCully CL, Godwin KS, Poplack DG. Methotrexate pharmacokinetics following administration of recombinant carboxypeptidase-G2 in rhesus monkeys. J Clin Oncol. 1992 Aug;10(8):1359-64. doi: 10.1200/JCO.1992.10.8.1359. PMID 1634927
- [Background] Widemann BC, Hetherington ML, Murphy RF, Balis FM, Adamson PC. Carboxypeptidase-G2 rescue in a patient with high dose methotrexate-induced nephrotoxicity. Cancer. 1995 Aug 1;76(3):521-6. doi: 10.1002/1097-0142(19950801)76:33.0.co;2-m. PMID 8625136
- [Background] Widemann BC, Balis FM, Murphy RF, Sorensen JM, Montello MJ, O'Brien M, Adamson PC. Carboxypeptidase-G2, thymidine, and leucovorin rescue in cancer patients with methotrexate-induced renal dysfunction. J Clin Oncol. 1997 May;15(5):2125-34. doi: 10.1200/JCO.1997.15.5.2125. PMID 9164227